CLINICAL TRIAL: NCT04434989
Title: Stereotactic Body Radiotherapy Versus Ablation for Perivascular Hepatocellular Carcinoma: A Phase 2, Multicenter, Randomized Controlled Trial
Brief Title: SBRT Versus Ablation for Perivascular Hepatocellular Carcinoma
Acronym: SAIL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Ming Kuang, Vice President, First Affiliated Hospital, Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HCC2020
Record Dates: First submitted 2020-06-15; First posted 2020-06-17 (Actual); Last update posted 2020-06-17 (Actual); Status verified 2020-06

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Radiosurgery; Radiofrequency Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stereotactic Body Radiation Therapy (Experimental): SBRT is defined as a special radiotherapy technique. The high dose of radiotherapy is accurately injected into the tumor lesion in one to several times using external irradiation technique. Then the tumor is exposed to high dose and the surrounding normal tissue to low dose.
  Interventions: Radiation: Stereotactic Body Radiation Therapy
- Radiofrequency Ablation (Active Comparator): Percutaneous radiofrequency ablation to the tumor
  Interventions: Procedure: radiofrequency ablation

INTERVENTIONS:
Radiation: Stereotactic Body Radiation Therapy — SBRT for perivascular HCC
  Other Names: SBRT
  Arms: Stereotactic Body Radiation Therapy
Procedure: radiofrequency ablation — RFA for perivascular HCC
  Other Names: RFA
  Arms: Radiofrequency Ablation

SUMMARY:
This trial is a multi-center, phase III, randomized (1:1) clinical trial. The aim is to explore the efficacy and safety of SBRT for perivascular hepatocellular carcinoma, compared with RFA.

DETAILED DESCRIPTION:
The primary endpoint is 1-year local recurrence rate and disease-free survival. We planned to recruit 170 patients who diagnosed as perivascular hepatocellular carcinoma. The patients will be randomized into SBRT group and RFA group as 1:1 ratio.

ELIGIBILITY:
Inclusion Criteria:

1. Primary hepatocellular carcinoma or recurrent hepatocellular carcinoma after curative treatment.
2. Unifocal tumor ≤5cm
3. Closed to great vessels (diameter ≥3mm)
4. ECOG score 0-1
5. Child-Pugh grade A or B7
6. Sufficient liver and kidney function

Exclusion Criteria:

1. Vascular invasion
2. Extra-hepatic metastasis
3. Received TACE before
4. Inflammation of local skin
5. Dysfunction of liver, kidney or bone marrow.
6. Concomitant other malignant tumor or HIV infection

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
1-year local recurrence rate | 1 year
  The rate of participants who have recurrence in treating area in 1 year to all the participants
Disease-free survival | 2 years
  The duration between radomization and recurrence, progression or death

SECONDARY OUTCOMES:
Overall survival | 2 years
  The duration between radomization and death
2-year recurrence rate | 2 years
  The rate of participants who have recurrence in 2 years to all the participants
Adverse events | 2 years
  The incidence rate of severe adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Kang TW, Lim HK, Lee MW, Kim YS, Choi D, Rhim H. Perivascular versus nonperivascular small HCC treated with percutaneous RF ablation: retrospective comparison of long-term therapeutic outcomes. Radiology. 2014 Mar;270(3):888-99. doi: 10.1148/radiol.13130753. Epub 2013 Nov 22. PMID 24475820
- [Background] Kim N, Cheng J, Jung I, Liang J, Shih YL, Huang WY, Kimura T, Lee VHF, Zeng ZC, Zhenggan R, Kay CS, Heo SJ, Won JY, Seong J. Stereotactic body radiation therapy vs. radiofrequency ablation in Asian patients with hepatocellular carcinoma. J Hepatol. 2020 Jul;73(1):121-129. doi: 10.1016/j.jhep.2020.03.005. Epub 2020 Mar 10. PMID 32165253
- [Background] Wahl DR, Stenmark MH, Tao Y, Pollom EL, Caoili EM, Lawrence TS, Schipper MJ, Feng M. Outcomes After Stereotactic Body Radiotherapy or Radiofrequency Ablation for Hepatocellular Carcinoma. J Clin Oncol. 2016 Feb 10;34(5):452-9. doi: 10.1200/JCO.2015.61.4925. Epub 2015 Nov 30. PMID 26628466
- [Background] Rajyaguru DJ, Borgert AJ, Smith AL, Thomes RM, Conway PD, Halfdanarson TR, Truty MJ, Kurup AN, Go RS. Radiofrequency Ablation Versus Stereotactic Body Radiotherapy for Localized Hepatocellular Carcinoma in Nonsurgically Managed Patients: Analysis of the National Cancer Database. J Clin Oncol. 2018 Feb 20;36(6):600-608. doi: 10.1200/JCO.2017.75.3228. Epub 2018 Jan 12. PMID 29328861